CLINICAL TRIAL: NCT07313709
Title: Measuring the Feasibility and Effect of a Virtual Reality Cognitive Training Intervention for Brain Cancer Survivors.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Anthony Faiola, Principal Investigator, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UCCC-BN-25-01
Record Dates: First submitted 2025-10-29; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-10

CONDITIONS: Brain Cancer
Keywords: virtual reality; cognitive impairment; brain cancer; cancer survivorship; non-invasive therapeutic medicine
MeSH Terms: conditions — Brain Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: After eligibility is confirmed, participants will be randomized into either the Experimental (Virtual Reality) or Control (Word Search Puzzles) Arms. Participants will be randomized in blocks of 4 through a computer-generated randomization such that the final n in the experimental arm is 20 and the control arm is 20. If a participant has to drop out of the study for any reason after randomization and start of the baseline/onboarding phase (e.g., due to motion sickness during participation) this will be considered in the assessment of feasibility for this study and they will not be replaced. The UCCC Data Manager will issue subject randomization to the study team upon receipt of confirmation of eligibility (with eligibility being confirmed per UCCC CTO workflows).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Virtual Reality - VR) (Experimental): Experimental (VR) Participants ONLY:
  Participants randomized to using Virtual Reality-Cognitive Rehab Training (VR-CRT) will have the game already installed/uploaded in the VR headset and ready for use, with their pre-determined participant number for user login and password assigned.
  Interventions: Other: Virtual Reality System
- Control (WSP) (Active Comparator): Control (WSP) Participants ONLY:
  Participants randomized to the control group will have their WSP packet with pre-selected word puzzles that provide a cognitive stimulus but without an increase in complexity. The instructions provided will state how participants should complete the WSP day-by-day. The dated completed WSPs, along with weekly check-ins by the study CRC will constitute the record for the participant's progress over four weeks. CRCs will notify the PI via email if during the call the participant indicates they have missed any of the WSPs during a given week.
  Interventions: Other: Word Search Puzzles

INTERVENTIONS:
Other: Virtual Reality System — Participants randomized to using VR-CRT will have the game already installed/uploaded in the VR headset and ready for use, with their pre-determined participant number for user login and password assigned.
  Arms: Experimental (Virtual Reality - VR)
Other: Word Search Puzzles — Participants randomized to the control group will have their WSP packet with pre-selected word puzzles that provide a cognitive stimulus but without an increase in complexity. The instructions provided will state how participants should complete the WSP day-by-day. The dated completed WSPs, along with weekly check-ins by the study CRC will constitute the record for the participant's progress over four weeks. CRCs will notify the PI via email if during the call the participant indicates they have missed any of the WSPs during a given week.
  Arms: Control (WSP)

SUMMARY:
The study is focused on assessing the feasibility and effect of a virtual reality training intervention for improving the survivorship journey of brain cancer survivors, post-treatment. The gaming intervention is intended to reduce cognitive impairment, while increasing well-being, mental health, and quality of life.

DETAILED DESCRIPTION:
This study is focused on assessing the feasibility, acceptability and effect of a virtual reality training intervention for improving the survivorship journey of brain cancer survivors, post-treatment. The gaming intervention is intended to reduce cognitive impairment, while increasing well-being, mental health, and quality of life. In sum, the potential impact of this research is to realize the capability of virtual reality cognitive rehabilitation training (VR-CRT) by mitigating brain cancer survivors (BCS) cognitive decline, while improving overall quality of life (QOL).

ELIGIBILITY:
Inclusion Criteria:

1. Low grade glioma survivors.
2. Have mild cognitive impairment (MCI) per MoCA (defined as any score between 18 and 25).
3. Completed all cancer treatment for their low-grade glioma (including chemotherapy, immunotherapy, radiation therapy and surgical procedures) and are now >30 days to 24 months from the date of last treatment.
4. Age 18 years or older.
5. English speaking.
6. Able to provide consent without use of a Legally Authorized Representative
7. Available to play the VR game or complete word search puzzles once per day for six days per week for four consecutive weeks in their home (per patient self-report).
8. Have a reliable phone number by which they can be reached to make arrangement for testing and for follow-up calls.

Exclusion Criteria:

* 1. History of serious mental or severe psychiatric illnesses (e.g., bi-polar disorder, schizophrenia etc....).

  a. Note: Anxiety or depression are not exclusionary. 2. History or known neurodegenerative diseases such as Alzheimer's disease, vascular dementia or any other form of advanced neurodegenerative or neuro-cognitive diseases.

  3. History of drug intoxication/overdose (addiction history). 4. History of acute traumatic brain injury. 5. History of stroke causing a cognitive deficit only. 6. Vision impairments including legal blindness.

  a. Note: patients with corrected vision (e.g., glasses or contacts) or who are color-blind are eligible.

  7. Incarcerated at the time of study enrollment. 8. Enrolled in another clinical trial which does not permit co-enrollment. 9. Any medical condition precluding safe use of VR headset and hand control technology, including patients with medical devices, including cardiac pacemakers, hearing aids/cochlear implants and defibrillators.

  10. History of motion sickness per patient self-report.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility defined as >80% (> 16 participants out of 20) able to complete the experimental arm study in 4 weeks. | 4 weeks
  FEASIBILITY: Measure the feasibility of using VR-CRT and Control (i.e., paper-based Word-search puzzles (WSP)) with brain cancer survivors (BCS) experiencing cancer-related cognitive impairment (CRCI).
  Feasibility: will be defined as >80% (> 16 participants out of 20) able to complete the experimental arm study in 4 weeks. Since the standard/control arm is well established and routine, feasibility evaluation is not required in this arm. (If subjects withdraw in disproportion in two arms after the randomization, the study may be suspended for further evaluation.)
Acceptability defined as scores of >8 on each subscale of the Senior Technology Acceptance Model (STAM).54 The STAM (Short Version) measures four attitudes towards technology on a Likert scale of 1-10. | 4 weeks
  ACCEPTABILITY: Measure the acceptability of using VR-CRT and Control (i.e., paper-based Word-search puzzles (WSP)) with brain cancer survivors (BCS) experiencing cancer-related cognitive impairment (CRCI). Acceptability: will be defined as scores of >8 on each subscale of the Senior Technology Acceptance Model (STAM).54 The STAM (Short Version) measures four attitudes towards technology on a Likert scale of 1-10. (See sections 3.1, 17.1 for detail.) This score of >8 for all 14 responses will be calculated as an average of all of the completed sub-scales per each subject. Any missing sub-scales (non-response by subjects) will not be considered into the calculation of the mean per subject. The score of >8 must be observed in >80% (>32 participants) to be considered acceptable.
Effect of VR-CRT (and Control) on cognitive function measured by scores at baseline and post-intervention,using 1.) Hopkins Verbal Learning Test | 4 weeks
  EFFECT: Estimate the effect of VR-CRT (and Control) on brain cancer survivors' cognitive function such as memory, attention/focus, processing speed, and executive function. Effect: will be measured by 1.) Hopkins Verbal Learning Test (HVLT)
Effect of VR-CRT (and Control) on cognitive function measured by scores at baseline and post-intervention,using 2.) Controlled Oral Word Association | 4 weeks
  EFFECT: Estimate the effect of VR-CRT (and Control) on brain cancer survivors' cognitive function such as memory, attention/focus, processing speed, and executive function. Effect: will be measured by comparing scores collected at baseline and post-intervention, (i.e., at the conclusion of a four-week intervention period) using 2.) Controlled Oral Word Association (COWA)
Effect of VR-CRT (and Control) on cognitive function measured by scores at baseline and post-intervention,using 3.) Trail Making A-B | 4 weeks
  EFFECT: Estimate the effect of VR-CRT (and Control) on brain cancer survivors' cognitive function such as memory, attention/focus, processing speed, and executive function. Effect: will be measured by comparing scores collected at baseline and post-intervention, (i.e., at the conclusion of a four-week intervention period) using 3.) Trail Making A-B (TMa/b).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided